CLINICAL TRIAL: NCT00770601
Title: A Multi-Center, Open Label, 24-Month Treatment Study to Establish the Safety, Tolerability, Efficacy, Pharmacokinetics of Canakinumab (Anti-IL-1 Beta Antibody) in Patients With NOMID / CINCA Syndrome
Brief Title: Canakinumab to Treat Neonatal-Onset Multisystem Inflammatory Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CACZ885D2201; 09-AR-0006 (Other: NIDDK-NIAMS IRB)
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Results first posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: NOMID; CINCA Syndrome
Keywords: NOMID; CINCA Syndrome; Canakinumab
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes | interventions — canakinumab

ARMS (1):
- Canakinumab (Experimental): Participants received body-weight stratified dosage of canakinumab treatment at 300 milligrams (mg) (for participants weighing more than 40 kilograms (kg)) and at 2 mg/kg (for participants weight less than or equal to 40 kg) subcutaneously every 4-8 weeks as per investigator discretion for a treatment period of 6 months. The first 3 Neonatal-Onset Multisystem Inflammatory Disease (NOMID) participants enrolled received a dose of 150 mg (>40 kg) and 2 mg/kg for children <40 kg. Since this dose was insufficient to fully control the symptoms of the disease the 300 mg / 4mg/kg dose was introduced by Protocol Amendment 2.
  Interventions: Drug: Canakinumab

INTERVENTIONS:
Drug: Canakinumab

SUMMARY:
This study will examine whether a medicine called canakinumab is safe and effective for treating patients with neonatal-onset multisystem inflammatory disease (NOMID), also known as chronic infantile neurologic, cutaneous, articular (CINCA) syndrome. This disease can cause rash, joint deformities, brain inflammation, problems with the eyes and learning difficulties. Canakinumab is an experimental drug that inhibits the action of a protein produced by the body called human IL-1beta, which is responsible for the symptoms in NOMID and also contributes to many other kinds of inflammatory diseases.

Patients 2 years of age and older with NOMID / CINCA may be eligible for this study. Participants undergo the following procedures:

Screening Phase

* Medical history and review of medical records
* Blood tests
* Daily diary of symptoms and medicines take

Washout/Lead-in Phase

* Discontinuation of anakinra or other medications, a 6 to 48-hour run-in period (only for patients who discontinued anakinra or other IL-1 blocking therapy).

Treatment Phase

* Injection of canakinumab under the skin every 8 weeks for 6 months
* Monitoring and evaluations during treatment, including:
* Quality-of-life questionnaires and daily diary
* Vital signs measurements (heartbeat, blood pressure, temperature)
* Blood tests
* Electrocardiogram
* Tuberculosis skin test
* Neurological, eye and skin examinations at beginning and end of study
* Cognitive evaluation at beginning and end of study
* Lumbar puncture (spinal tap) at the beginning of the study, 2 weeks after the second dosing of canakinumab and at the end of the study
* X-rays and bone density scan at beginning and end of study
* Magnetic resonance imaging (MRI) of the head at beginning and end of study

Follow-up Phase

* Monthly clinic visits after the last dose of canakinumab for a minimum of 60 days

End-of-Study Evaluation

* Series of tests 8 weeks after last dose of canakinumab to evaluate treatment response and side effects

DETAILED DESCRIPTION:
This open-label study was designed to investigate the safety, tolerability, efficacy, pharmacokinetics and pharmacodynamics of canakinumab, a fully human anti-interleukin-1beta (anti-IL-1beta) monoclonal antibody, in patients with NOMID / CINCA syndrome. A total of 25 to 30 patients will be enrolled into the study. The study consists of two stages:

In the first pilot stage it is planned to enroll 5 patients undergoing PK/PD assessments in blood and cerebrospinal fluid (CSF), and monitoring of efficacy (CNS relapse and inflammatory relapse) to confirm the dose and dosing regimen before enlarging the number of patients enrolled into the study. Up to 5 additional patients may be enrolled in this stage if the variability of the responses to treatment is high. Interim analyses will be conducted as required. Following Stage 1, a second confirmatory stage will be conducted, enrolling 20 additional patients. In this stage patients will be treated with the dose and dosing regimen based on the assessment of the efficacy profile in Stage 1 and exploratory PK/PD assessment. In each stage there will be a 3-week screening period to collect pre-treatment parameters, a run-in period (only for patients who discontinue anakinra), a baseline evaluation prior to each drug administration, a 24-week treatment period with fixed dosing of canakinumab, and a study completion visit. Patients whose body weight is greater than 40 kg will receive canakinumab 150 mg as a subcutaneous (s.c.) injection, and patients with a body weight less than or equal to 40 kg will receive canakinumab 2 mg/kg s.c. Patients will be administered canakinumab every 8 weeks and will undergo an observation period after each dose administration in order to evaluate the response to treatment. Patients who do not achieve complete remission following canakinumab injection in any treatment period will be re-dosed within Day 15 or receive the following dose adjustments:

* 300 mg s.c. (or 4 mg/kg for patients with a body weight less than or equal to 40 kg)
* 450 mg s.c. (or 6 mg/kg for patients with a body weight less than or equal to 40 kg)
* 600 mg s.c. (or 8 mg/kg for patients with a body weight less than or equal to 40 kg)

End of Study will occur when patients discontinue from the study or complete this study. The End of Study visit should occur 8 weeks (plus or minus 1 week) after the last injection. All patients who complete the 6-month evaluation may be offered to enter an extension study (CACZ885D2201E1) conducted to assess long term safety and efficacy data.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Male and female patients of greater than or equal to 2 years of age at the time of the screening visit.
2. Patient's informed consent (for greater than or equal to 18 years of age), or in pediatric patients, parents' or legal guardian's informed consent and patient's assent to the protocol whenever possible.
3. Females of childbearing potential (young women who have had at least one menstrual period regardless of age) and/or aged greater than or equal to 8 years must have a negative serum pregnancy test at screening and a negative urine pregnancy test at each baseline prior to performance of any radiologic procedure or administration of study medication.
4. Women of childbearing age and men able to father a child, who are sexually active, must agree to use a form of effective method of contraception (e.g. birth control pills, abstinence, double-barrier contraception, etc.) during the study (from the date of screening) and for at least 3 months following the last dose. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
5. Presence, or history (prior to anakinra treatment), of at least 2 of the following clinical manifestations:

   * Typical NOMID urticarial rash.
   * Central nervous system (CNS) involvement: increased intracranial pressure (greater than 180 mm water), papilledema, cerebral spinal fluid pleocytosis (white cell count greater than 6 cells/mm(3)), stroke, seizures, and/or sensorineural hearing loss.
   * Typical arthropathic changes on X-rays: epiphysial and/or patellar overgrowth.
6. Onset of NOMID/CINCA before or at 6 months of age.
7. Patients requiring oral steroids, NSAIDs and/or disease-modifying antirheumatic drugs (DMARDs) can be enrolled if they are on a stable dose (oral steroids: less than 20 mg/day or less than or equal to 0.4 mg/kg prednisone or prednisone equivalent, whichever applies) for at least 4 weeks prior to the screening visit. Steroid therapy may be tapered during treatment with canakinumab after the first canakinumab treatment period / cycle, at the discretion of the investigator.
8. Negative tuberculin skin test reaction (PPD 5 tuberculin units or as according to local standard practice) (less than 5mm induration) at 48 to 72 hours after administration at the screening visit or within 2 months prior to the screening visit, according to national guidelines. Patients who have a positive PPD skin test with a documentation of BCG vaccination, who are at low environmental risk for tuberculosis (TB) infection or reactivation, and have a negative chest X-ray can be included. A positive PPD test will be defined using the MMWR 2000 guidance, summarized as criteria for tuberculin positivity by risk group.
9. Able to comply with the requirements of the study.

EXCLUSION CRITERIA:

Subjects meeting any of the following criteria will be excluded from entry into or continuation in the study unless sponsor approval is obtained:

1. Pregnant or breastfeeding women.
2. Participation in any clinical trial investigation within 4 weeks prior to dosing or longer if required by local regulation, with the exception of trials with anakinra and/or canakinumab.
3. In case of previous treatment with biologic agents or DMARDs, an appropriate washout period (as according to the recognized duration of effect and half lives) will be required for such patients to be eligible to participate in the trial, e.g.:

   Previous treatment and required washout period prior to baseline and thereafter:
   * Rituximab, 26 weeks
   * Infliximab, 12 weeks
   * Adalimumab, 8 weeks
   * Etanercept, 4 weeks
   * Anakinra, 1 day
   * Any other investigational biologics, 8 weeks
   * Leflunomide, 4 weeks
   * Thalidomide, 4 weeks
   * Cyclosporine, 4 weeks
   * i.v. immunoglobulin (i.v. Ig), 8 weeks
   * Dapsone, mycophenolate mofetil, 3 weeks
   * Corticosteroids greater than or equal to 20 mg/day or greater than 0.4 mg/kg prednisone or prednisone equivalent, whichever applies, 1 week
4. Donation or loss of 300 mL or more of blood within 8 weeks prior to dosing.
5. A past medical history of clinically significant ECG abnormalities or a family history of a prolonged QT-interval syndrome.
6. History of immunocompromise.
7. Positive test for or prior history of HIV (ELISA and Western blot), Hepatitis B (Hepatitis B surface antigen) or Hepatitis C.
8. Presence of active infections or a history of pulmonary TB infection with or without documented adequate therapy. Subjects with current active TB, or recent close exposure to an individual with active TB are excluded from the study.
9. Presence of any additional rheumatic disease or significant systemic disease. For example, major chronic infectious/ inflammatory/ immunologic disease (such as inflammatory bowel disease, psoriatic arthritis, spondyloarthropathy, systemic lupus erythematosus in addition to the autoinflammatory disease).
10. Treatment with a live virus vaccine during 3 months prior to baseline visit. No live vaccines will be allowed throughout the course of this study and up to 3 months following the last dose.
11. History of renal transplant.
12. History of malignancy. Subjects deemed cured of superficial malignancies such as cutaneous basal or squamous cell carcinomas, or in situ cervical cancer may be enrolled.
13. Presence of any of the following laboratory abnormalities: ALT or AST greater than 2 times the upper limit of normal (ULN), platelet count less than 100x10(9)/L.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2009-01-26 (Actual); Primary Completion 2011-02-17 (Actual); Study Completion 2011-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS), 9, Bethesda, Maryland, United States

REFERENCES:
- [Background] Goldbach-Mansky R, Dailey NJ, Canna SW, Gelabert A, Jones J, Rubin BI, Kim HJ, Brewer C, Zalewski C, Wiggs E, Hill S, Turner ML, Karp BI, Aksentijevich I, Pucino F, Penzak SR, Haverkamp MH, Stein L, Adams BS, Moore TL, Fuhlbrigge RC, Shaham B, Jarvis JN, O'Neil K, Vehe RK, Beitz LO, Gardner G, Hannan WP, Warren RW, Horn W, Cole JL, Paul SM, Hawkins PN, Pham TH, Snyder C, Wesley RA, Hoffmann SC, Holland SM, Butman JA, Kastner DL. Neonatal-onset multisystem inflammatory disease responsive to interleukin-1beta inhibition. N Engl J Med. 2006 Aug 10;355(6):581-92. doi: 10.1056/NEJMoa055137. PMID 16899778
- [Background] Hawkins PN, Lachmann HJ, Aganna E, McDermott MF. Spectrum of clinical features in Muckle-Wells syndrome and response to anakinra. Arthritis Rheum. 2004 Feb;50(2):607-12. doi: 10.1002/art.20033. PMID 14872505
- [Background] Hirsch E, Irikura VM, Paul SM, Hirsh D. Functions of interleukin 1 receptor antagonist in gene knockout and overproducing mice. Proc Natl Acad Sci U S A. 1996 Oct 1;93(20):11008-13. doi: 10.1073/pnas.93.20.11008. PMID 8855299
- [Derived] Sibley CH, Chioato A, Felix S, Colin L, Chakraborty A, Plass N, Rodriguez-Smith J, Brewer C, King K, Zalewski C, Kim HJ, Bishop R, Abrams K, Stone D, Chapelle D, Kost B, Snyder C, Butman JA, Wesley R, Goldbach-Mansky R. A 24-month open-label study of canakinumab in neonatal-onset multisystem inflammatory disease. Ann Rheum Dis. 2015 Sep;74(9):1714-9. doi: 10.1136/annrheumdis-2013-204877. Epub 2014 Jun 6. PMID 24906637
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/A_2009-AR-0006.html
- See also: link to the results on Novartis results database — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=5464

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at a single center in United States
Pre-assignment Details: A total of 7 participants were screened of which only 6 participants were randomized into the study, as one participant withdrew consent before dosing.
Groups:
- Canakinumab (ACZ885): Participants received body-weight stratified dosage of canakinumab treatment at 300 milligrams (mg) (for participants weighing more than 40 kilograms (kg)) and at 2 mg/kg (for participants weight less than or equal to 40 kg) subcutaneously every 4-8 weeks as per investigator discretion for a treatment period of 6 months. The first 3 Neonatal-Onset Multisystem Inflammatory Disease (NOMID) participants enrolled received a dose of 150 mg (>40 kg) and 2 mg/kg for children <40 kg. Since this dose was insufficient to fully control the symptoms of the disease the 300 mg / 4mg/kg dose was introduced by Protocol Amendment 2.
Period: Overall Study
Arm/Group | Canakinumab (ACZ885)
Started | 7
Completed | 6
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The analysis was performed on all participants randomized and received at least on dose of study drug.
Groups:
- Canakinumab (ACZ885): Participants received body-weight stratified dosage of canakinumab treatment at 300 mg (for participants weighing more than 40 kg) and at 2 mg/kg (for participants weight less than or equal to 40 kg) subcutaneously every 4-8 weeks as per investigator discretion for a treatment period of 6 months. The first 3 NOMID participants enrolled received a dose of 150 mg (>40 kg) and 2 mg/kg for children <40 kg. Since this dose was insufficient to fully control the symptoms of the disease the 300 mg / 4mg/kg dose was introduced by Protocol Amendment 2.
Arm/Group | Canakinumab (ACZ885)
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.7 (8.09)
Age, Customized [Count of Participants; unit: Participants]
  Children (2-11 years) | 1
  Adolescents (12-17 years) | 3
  Adults (18-64 years) | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 4
  Black | 1
  Asian | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 1
  Japanese | 1
  Mixed Ethinicity | 2
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Remission and Relapse After 6 Months of Canakinumab Treatment.
Description: The primary endpoint of the study was the percentage of participants experiencing a relapse Central nervous system (CNS) relapse and/or inflammatory relapse) during 6-month open label administration of canakinumab in participant with NOMID/Chronic Infantile Neurological, Cutaneous, Articular Syndrome (CINCA). Complete remission consisted of inflammatory remission and CNS remission. 1 Inflammatory (systemic) remission was defined as follows (all criteria to be fulfilled): -Serum C-reactive protein (CRP) AND serum amyloid A (SAA) ≤ 10 milligrams/litre AND -daily diary score (mean score/week) ≤ 2. 2) CNS remission was defined as follows: Headache score (from the daily diary, mean score/week) < 0.5 AND, when a lumbar puncture was performed: Normal values of white cell count (WBC) (≤15 cells/mm3) in CSF.
Time Frame: 6 months
Population: The primary analysis was performed on all participants randomized and received at least one dose of study drug. No participant was in stable full remission state as defined by the protocol.
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab (ACZ885)
Number analyzed (Participants) | 6
Percentage of participants | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV) for approx. 2 years
Arm/Group | Canakinumab (ACZ885)
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab (ACZ885) (N=6)
Staphylococcal infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab (ACZ885) (N=6)
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Ear pain (Ear and labyrinth disorders) | 2
Conjunctivitis allergic (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Condition aggravated (General disorders) | 1
Pyrexia (General disorders) | 2
Ear infection (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Joint injury (Injury, poisoning and procedural complications) | 2
Procedural pain (Injury, poisoning and procedural complications) | 1
Basophil count increased (Investigations) | 2
Blood albumin decreased (Investigations) | 1
Blood albumin increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood chloride increased (Investigations) | 1
Blood creatine phosphokinase decreased (Investigations) | 3
Blood creatine phosphokinase increased (Investigations) | 1
Blood creatinine decreased (Investigations) | 5
Blood glucose increased (Investigations) | 1
Blood triglycerides increased (Investigations) | 1
Blood uric acid decreased (Investigations) | 2
C-reactive protein increased (Investigations) | 3
CSF neutrophil count increased (Investigations) | 5
CSF protein increased (Investigations) | 4
CSF white blood cell count increased (Investigations) | 5
Eosinophil count increased (Investigations) | 3
Haematocrit decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Heart rate increased (Investigations) | 1
High density lipoprotein decreased (Investigations) | 1
Lymphocyte count increased (Investigations) | 2
Monocyte count increased (Investigations) | 1
Neutrophil count increased (Investigations) | 2
Platelet count decreased (Investigations) | 1
Platelet count increased (Investigations) | 1
Red blood cell count increased (Investigations) | 1
Red blood cell sedimentation rate increased (Investigations) | 2
White blood cell count increased (Investigations) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Costochondritis (Musculoskeletal and connective tissue disorders) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 4
Memory impairment (Nervous system disorders) | 1
Sinus headache (Nervous system disorders) | 1
Amenorrhoea (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Study was terminated prematurely due to multiple protocol amendments for change in study design; limited number of participants; availability of sufficient clinical data for higher doses of drug and lack of severe NOMID subjects for further evaluation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.